CLINICAL TRIAL: NCT07104175
Title: Value Analysis of Preoperative Nutritional Risk Screening 2002 (NRS2002) and Global Leadership Initiative on Malnutrition (GLIM) Screening in Predicting Postoperative Complications in Patients With Gastrointestinal Malignancies
Brief Title: Predictive Value of NRS2002 and GLIM for Complications After GI Malignancy Surgery
Status: Completed | Type: Observational
Sponsor: Third central hospital of Tianjin affiliated Nankai university (Network)
Responsible Party: Principal Investigator, Dongping Xu, Principal investigator, Third central hospital of Tianjin affiliated Nankai university
Other Study IDs: SZX-IRB-SOP-016(F)-002-01
Record Dates: First submitted 2025-07-27; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal Malignancies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Nutritional Risk Group (NRS2002 ≥ 3): Patients identified as being at nutritional risk based on the Nutritional Risk Screening 2002 (NRS2002) score (total score ≥ 3), assessed preoperatively within 24 hours of admission. These patients were followed to assess for postoperative outcomes.
- No Nutritional Risk Group (NRS2002 < 3): Patients identified as not being at significant nutritional risk based on the NRS2002 score (total score < 3), assessed preoperatively within 24 hours of admission. These patients served as the control group for the NRS2002 exposure and were followed to assess for postoperative outcomes.
- Malnutrition Group (GLIM Criteria): Patients diagnosed with malnutrition based on the Global Leadership Initiative on Malnutrition (GLIM) criteria, requiring at least one phenotypic and one etiologic criterion. Assessment was performed preoperatively within 24 hours of admission. Patients were followed to assess for postoperative outcomes. This group was also sub-categorized into moderate and severe malnutrition.
- No Malnutrition Group (GLIM Criteria): Patients who did not meet the GLIM criteria for malnutrition. Assessment was performed preoperatively within 24 hours of admission. These patients served as the control group for the GLIM exposure and were followed to assess for postoperative outcomes.

SUMMARY:
This prospective cohort study investigates and compares the predictive power of two nutritional assessment tools, the Nutritional Risk Screening 2002 (NRS2002) and the Global Leadership Initiative on Malnutrition (GLIM) criteria. The study aims to determine how well these tools can predict postoperative complications in patients with gastrointestinal malignancies who are undergoing surgical resection.

DETAILED DESCRIPTION:
Malnutrition is a common and severe problem in patients with gastrointestinal (GI) malignancies, adversely affecting surgical outcomes. This prospective cohort study was designed to evaluate and compare the predictive utility of two key nutritional assessment tools. Patients scheduled for elective curative-intent surgery for GI malignancies were enrolled. Within 24 hours of admission, each patient's nutritional status was assessed using both the Nutritional Risk Screening 2002 (NRS2002) and the Global Leadership Initiative on Malnutrition (GLIM) criteria. The study followed these patients through their hospital stay and post-discharge to collect data on the primary outcome of postoperative complications, as well as secondary outcomes including length of hospital stay, hospitalization costs, and unplanned 30-day and 60-day readmissions. The objective is to provide evidence to guide clinicians in using NRS2002 and GLIM for preoperative risk stratification and to identify patients who may benefit from nutritional interventions to improve surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histopathologically confirmed primary gastrointestinal malignancy (e.g., esophageal, gastric, colorectal cancer).
* Planned curative-intent surgical resection.
* No prior anti-tumor treatments such as surgery, radiotherapy, chemotherapy, or immunotherapy for the current malignancy.
* Provision of written informed consent to participate in the study.

Exclusion Criteria:

* Presence of other concurrent systemic malignant tumors.
* Emergency surgery.
* Hospital stay less than 48 hours post-surgery.
* Incomplete critical clinical or nutritional data.
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥18 years) with a new, histopathologically confirmed diagnosis of a primary gastrointestinal malignancy (e.g., esophageal, gastric, colorectal cancer). These patients were admitted to a single tertiary care center for elective, curative-intent surgical resection between December 2019 and December 2024. The population represents individuals who had not received prior anti-tumor treatments for their current malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Complications | Up to 30 days post-surgery
  Measured as the number of patients experiencing one or more postoperative complications. Complications were defined and graded according to the Clavien-Dindo classification system and the "Expert Consensus on Postoperative Complications Registration for Gastrointestinal Tumor Surgery (2018 Edition)". Major complications were defined as Clavien-Dindo grade III or higher.

SECONDARY OUTCOMES:
Length of Hospital Stay | Up to 60 days post-surgery (data collected at discharge)
  The total duration of the index hospitalization, measured from the date of admission to the date of discharge.
Intensive Care Unit (ICU) Admission Rate | Up to 30 days post-surgery
  The percentage of patients admitted to the ICU at any point during their postoperative hospital stay.
Unplanned 30-Day Readmission Rate | Within 30 days of discharge
  The percentage of patients who had an unplanned hospital readmission for any reason.
Unplanned 60-Day Readmission Rate | Within 60 days of discharge
  The percentage of patients who had an unplanned hospital readmission for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Central Hospital of Tianjin, Tianjin, Tianjin Municipality, China